CLINICAL TRIAL: NCT00461838
Title: Outcome After Multidisciplinary CO2 Laser Laparoscopic Excision of Deep Infiltrating Colorectal Endometriosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Christel Meuleman, MD, University Hospitals Leuven
Other Study IDs: ML2818 - 22/10/2004
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Endometriosis
Keywords: colorectal endometriosis; deep infiltrating endometriosis; dysmenorroe; dyspareunia; quality of life
MeSH Terms: conditions — Endometriosis; Dyspareunia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Endometriosis was proven by histologic examination of excised lesions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All women (n=56) who had undergone CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with active involvement of colorectal surgeon and/or urologist were selected retrospectively from the list of all patients (n=more than 2000) operated at the Leuven University Fertility Centre (LUFc) between September 1996 and July 2004.
  Interventions: Procedure: multidisciplinary laparoscopy; Other: Questionnaires

INTERVENTIONS:
Procedure: multidisciplinary laparoscopy — Multidisciplinary (with active involvement of the colorectal surgeon/urologist) fertility-sparing CO2 laser laparoscopic radical excision of deep infiltrating endometriosis.
Other: Questionnaires — Patients (n=56) were asked to complete questionnaires regarding quality of life (QOL), pain, fertility and sexuality to compare their status before and after surgery, and their medical files were analyzed.

SUMMARY:
Improved pain, sexuality and quality of life, high fertility and low complication and recurrence rates after multidisciplinary CO2 laser laparoscopic excision of deep infiltrating colorectal endometriosis.

DETAILED DESCRIPTION:
All women (n=56) who had undergone CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with active involvement of colorectal surgeon and/or urologist were selected retrospectively from the list of all patients (n=more than 2000) operated at the Leuven University Fertility Centre (LUFc) between September 1996 and July 2004.

All 56 multidisciplinary operated patients were asked to complete the Oxford Endometriosis Quality of Life questionnaire, a sexual activity questionnaire and visual analogue scales (VAS) for dysmenorroe, chronic pelvic pain and deep dyspareunia, to compare their status before surgery and at the moment of the evaluation (January 2005).

ELIGIBILITY:
Inclusion Criteria:

* All women (n=56) who had undergone CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with active involvement of colorectal surgeon and/or urologist
* operated at the Leuven University Fertility Centre (LUFc) between September 1996 and July 2004

Exclusion Criteria:

* Women who had undergone CO2 laser laparoscopic excision of deep infiltrating endometriosis without active involvement of colorectal surgeon and/or urologist

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women (n=56) who had undergone CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with active involvement of colorectal surgeon and/or urologist were selected retrospectively from the list of all patients (n=more than 2000) operated at the Leuven University Fertility Centre (LUFc) between September 1996 and July 2004.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 1996-09; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
complication rate, cumulative recurrence and cumulative fertility rate, pain, quality of life and sexual satisfaction | median follow-up: 29 months (range 6 - 76 months)

CONTACTS AND LOCATIONS:
Overall Officials: Christel LC Meuleman, MD, Principal Investigator — University Hospital Gasthuisberg, Catholic University, Leuven, Belgium; Thomas D'Hooghe, MD, PhD, Study Director — University Hospital Gasthuisberg, Catholic University, Leuven, Belgium
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium